CLINICAL TRIAL: NCT00565968
Title: A Phase I Dose Escalation Trial to Evaluate Safety and Efficacy of Oral Sorafenib (Nexavar) With Regional Melphalan Via Normothermic Isolated Limb Infusion (ILI) in Patients With Intransit Extremity Melanoma
Brief Title: Sorafenib and Isolated Limb Infusion of Melphalan in Treating Patients With Stage III Melanoma of the Arm or Leg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001344; CDR0000575427
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Melanoma (Skin)
Keywords: stage IIIB melanoma; stage IIIC melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Melphalan; Sorafenib; Gene Expression Profiling; Blotting, Western

ARMS (1):
- Sorafenib dose escalation (Experimental)
  Interventions: Drug: melphalan; Drug: sorafenib tosylate; Genetic: gene expression analysis; Genetic: protein expression analysis; Genetic: western blotting; Other: pharmacological study

INTERVENTIONS:
Drug: melphalan
Drug: sorafenib tosylate
Genetic: gene expression analysis
Genetic: protein expression analysis
Genetic: western blotting
Other: pharmacological study

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sorafenib may also make tumor cells more sensitive to melphalan. Giving sorafenib together with an isolated limb infusion of melphalan may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of sorafenib when given together with an isolated limb infusion of melphalan in treating patients with stage III melanoma of the arm or leg.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the dose-limiting toxicities and maximum tolerate dose of systemic sorafenib tosylate in combination with regionally administered melphalan by isolated limb infusion in patients with stage IIIB or IIIC intransit extremity melanoma.

Secondary

* To characterize the safety and tolerability of this regimen in these patients.
* To assess the antitumor activity of this regimen, as evidenced by best overall response and duration of response, in these patients.
* To characterize the duration of progression-free survival of these patients.
* To characterize the pharmacokinetics of melphalan.
* To assess alterations in selected gene and protein expression profiles following treatment.

OUTLINE: This is a multicenter, dose-escalation study of sorafenib tosylate.

Patients receive oral sorafenib tosylate twice daily on days 1-14 and melphalan via isolated limb infusion into the upper or lower extremities on day 8.

Patients undergo tumor biopsies at baseline and in weeks 2 and 12 for gene expression analysis and western blot analysis. Patients also undergo blood sample collection periodically for pharmacokinetic analysis of melphalan.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary or recurrent extremity melanoma

  * Stage IIIB or IIIC disease

    * Patients with stage IIIC disease must have had regional lymph nodes previously removed
* Disease to be treated by regional therapy must be distal to the planned site of tourniquet placement
* Bidimensionally measurable disease by caliper or radiological method

  * Must have identifiable target lesions for disease assessment

    * Patients with a single lesion must have archived tumor tissue available for research analysis
* No stage IV disease
* No known brain metastasis

  * Patients with neurological symptoms must have undergone a CT scan or MRI of the brain within the past 4 weeks to exclude brain metastasis

PATIENT CHARACTERISTICS:

* ECOG or Zubrod performance status 0-1
* Life expectancy > 6 months
* Hemoglobin ≥ 9.0 g/dL
* WBC ≥ 3,000/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* ALT and AST ≤ 2.5 x ULN
* INR < 1.5 or PT/PTT normal
* Creatinine ≤ 1.5 x ULN
* Not pregnant or nursing
* Negative serum pregnancy test
* Fertile patients must use effective contraception
* Must have a palpable femoral or axillary pulse in the extremity to be treated
* No cardiac disease, including any of the following:

  * NYHA class III or IV congestive heart failure
  * Unstable angina (i.e., angina symptoms at rest) or new onset angina within the past 3 months
  * Myocardial infarction within the past 6 months
* No cardiac ventricular arrhythmias requiring antiarrhythmic therapy
* No uncontrolled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg or diastolic BP > 90 mm Hg, despite optimal medical management
* No known HIV infection
* No chronic hepatitis B or C
* No active clinically serious infection > CTCAE grade 2
* No thrombotic or embolic events (e.g., cerebrovascular accident or transient ischemic attacks) within the past 6 months
* No signs or symptoms of vascular insufficiency (i.e., any history of blood clots or other ischemic peripheral vascular disease)
* No evidence or history of bleeding diathesis or coagulopathy
* No pulmonary hemorrhage or bleeding event ≥ CTCAE grade 2 within the past 4 weeks
* No other hemorrhage or bleeding event ≥ CTCAE grade 3 within the past 4 weeks
* No serious nonhealing wound, ulcer, or bone fracture
* No significant traumatic injury within the past 4 weeks
* No condition that impairs the patient's ability to swallow whole pills
* No malabsorption problem
* No known history of allergic reactions and/or hypersensitivity to melphalan, sorafenib tosylate, or any other agent used in the study
* No psychiatric condition or diminished capacity that would compromise giving informed consent, or interfere with study compliance
* No history of other malignancies, except for any of the following:

  * Adequately treated basal cell or squamous cell carcinoma of the skin
  * Curatively treated in situ carcinoma of the uterine cervix, prostate cancer, or superficial bladder cancer
  * Other curatively treated solid tumor with no evidence of disease for ≥ 5 years

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* No prior sorafenib tosylate
* Prior melphalan via isolated limb infusion allowed
* No antineoplastic therapy, radiotherapy, or any other investigational drug within the past 4 weeks
* No major surgery or open biopsy within the past 4 weeks
* No concurrent Hypericum perforatum (St. John wort) or rifampin
* Concurrent anti-coagulation treatment with warfarin or heparin allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 1 year

SECONDARY OUTCOMES:
Safety and tolerability | 2 years
Antitumor activity, as evidenced by best overall response and duration of response | 3 years
Duration of progression-free survival | 3 years
Pharmacokinetics of melphalan | 3 years
Tumor gene and protein expression profiles following treatment | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S. Tyler, MD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States